CLINICAL TRIAL: NCT06921096
Title: Effect of Tai Chi Exercise and Its Cessation on Internet Addiction in College Students: A Randomized Controlled Trial
Brief Title: Cessation on Internet Addiction in College Students
Acronym: IAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu Sport University (Other)
Responsible Party: Principal Investigator, Cheng Liang, Director, Chengdu Sport University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Internet Addiction Disorder
Record Dates: First submitted 2025-03-29; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Internet Addiction Disorder
Keywords: Internet Addiction Disorder; Tai Chi
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Maintain your original lifestyle without engaging in regular physical exercise. Participants were contacted every two weeks via WeChat or in person to monitor their conditions and ensure no extra exercise or medication use.
- Tai Chi group (Experimental): The Tai Chi group practiced 24-form simplified Tai Chi for 12 weeks, 3 times/week, 60 minutes/session (including 5-minute warm-up and 5-minute cool-down) at our university's track, under professional coaching, from 8:00-9:10 AM. The first 4 weeks were for learning, and the next 8 for consolidation. Then, we will observe all participants for an additional 4 weeks (Week 16) as a follow-up.
  Interventions: Other: Tai Chi

INTERVENTIONS:
Other: Tai Chi — The Tai chi group practiced 24-form simplified Tai Chi for 12 weeks, 3 times/week, 60 minutes/session (including 5-minute warm-up and 5-minute cool-down) at our university's track, under professional coaching, from 8:00-9:10 AM. The first 4 weeks were for learning, and the next 8 for consolidation.
  Arms: Tai Chi group

SUMMARY:
This study aimed to explore the intervention effect of Tai Chi exercise on internet addiction in college students and its maintenance effect after cessation, providing a scientific basis for the application of Tai Chi in internet addiction intervention among college students. Fifty-one non-sports-major college students with mild or moderate internet addiction were randomly divided into a Tai Chi group (n = 23) and a control group (n = 24). The Tai Chi group underwent 12 weeks of Tai Chi exercise, while the control group maintained their regular study schedule without additional physical exercise. The Chinese Internet Addiction Scale and serum dopamine and β-Endorphin levels were assessed at baseline, week 12, and week 16.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-25;
* CIAS scores of 26-53 (low internet dependence), 54-80 (moderate dependence), or 81-104 (high dependence). Only mild and moderate cases were included;
* non-sports majors; the study followed the Declaration of Helsinki, and all participants understood the purpose and signed consent forms.

Exclusion Criteria:

* Severe IAD (CIAS score >80);
* Tai Chi practice within 6 months;
* regular exercise habits;
* history of depression/anxiety or undergoing psychological treatment;
* use of medications affecting mental state or neurotransmitter levels.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-16 (Estimated)

PRIMARY OUTCOMES:
Internet Addiction Scale Survey | 16 weeks
  The CIAS, tailored to Chinese college students' psychological traits, was used. It has 26 items across five dimensions: compulsive symptoms, withdrawal symptoms, tolerance symptoms, interpersonal and health problems, and time management problems. It's a 4-point self-report Likert scale (1="extremely disagree" to 4="extremely agree"). The scale has good reliability and validity, with factor consistency coefficients of 0.70-0.82 and internal consistency of 0.9446[21]. The total CIAS score is the sum of all items, with higher scores indicating greater dependence and addiction risk. The CIAS was administered at baseline, week 12, and week 16 for both groups.

SECONDARY OUTCOMES:
Serum Dopamine | 16 weeks
  At baseline, week 12, and week 16, 2 ml of fasting venous blood was collected from participants between 7:00-8:00 AM. Serum dopamine levels was measured using radioimmunoassay on a Beckman DXC800 autoanalyzer, with reagents from IBL (Germany). All steps followed the kit instructions, and absorbance was measured at 450 nm to calculate concentrations.
Serum β-Endorphin | 16 weeks
  At baseline, week 12, and week 16, 2 ml of fasting venous blood was collected from participants between 7:00-8:00 AM. Serum β-Endorphin levels was measured using radioimmunoassay on a Beckman DXC800 autoanalyzer, with reagents from IBL (Germany). All steps followed the kit instructions, and absorbance was measured at 450 nm to calculate concentrations.

IPD SHARING:
Plan to Share IPD: Yes